CLINICAL TRIAL: NCT03216135
Title: Microbiome Involvement With Barrett's Esophagus and Progression to Esophageal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ochsner Health System (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Virendra Joshi, MD, Ochsner Health System
Other Study IDs: 2017113
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-03

CONDITIONS: Barrett Esophagus; Esophageal Cancer
Keywords: Microbiome
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue of the esophagus. Bacterial genomic DNA to be extracted from tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- (GERD) with no Barrett's Esophagus: Squamous epithelium from patient with gastroesophageal reflux disease (GERD) with no BE or EAC diagnosed will be collected and a control sample (area with no disease).
- Barrett's Esophagus: BE/columnar epithelium from patient diagnosed with BE and a control sample (area with no disease).
- Cancer Tissue: Cancer tissue, and a control squamous epithelium from the same patient.

SUMMARY:
This study will examine the hypothesis that altered esophageal microbiome leads to the development of esophageal adenocarcinoma (EAC). The aims of the project are, firstly the confirmation of relational data on the study cohort, using the methods developed and applied at the laboratory at University of Queensland Diamantina Institute (UQDI). Second, to generate a tissue microarray resource future tissue in-situ validation of microbes. And finally, to develop a biobank of clinical isolates of relevant esophageal microbes for future functional studies.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease, GERD, can lead to a change of the esophagus lining to a protective cell type, termed Barrett's esophagus (BE). A diagnosis of BE greatly increases the risk of developing esophageal adenocarcinoma (EAC). The incidence of EAC has been rapidly rising in the last 30 years, and the cancer has a high mortality rate. Understanding the involvement of the esophageal microbiota could lead to prevention strategies to this increasing health concern.

This study will examine the hypothesis that altered esophageal microbiome leads to the development of esophageal adenocarcinoma (EAC). The aims of the project are, firstly the confirmation of relational data on the study cohort, using the methods developed and applied at the laboratory at University of Queensland Diamantina Institute (UQDI). Second, to generate a tissue microarray resource future tissue in-situ validation of microbes. And finally, to develop a biobank of clinical isolates of relevant esophageal microbes for future functional studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or females >18 years of age with known or suspected GERD, Barrett's Esophagus and or esophageal adenocarcinoma or from patients who have a history of either condition.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 10 samples of 3 specific tissue types (specified as the 3 groups) will be collected as well as control samples. The number of patients enrolled may vary due to the variance of tissue type per patient. Patients will be informed that the number of patients enrolled will depend on the number of tissues needed for the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-07-20 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Microbial community profiling | 9 months
  16S Ribosomal RNA (rRNA)gene sequencing

SECONDARY OUTCOMES:
Generate a tissue microarray | 9 months
  After retrieval of blocks, an experienced pathologist will mark the relevant tissue areas to process into microarray

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Health System, Kenner, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No